CLINICAL TRIAL: NCT00813267
Title: Mesenchymal Stem Cell Transplantation in the Treatment of Osteonecrosis of the Femoral Head
Brief Title: Mesenchymal Stem Cell for Osteonecrosis of the Femoral Head
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jianming Tan (Other)
Responsible Party: Sponsor-Investigator, Jianming Tan, Director, Fuzhou General Hospital
Organization: Fuzhou General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fuzhough1221
Record Dates: First submitted 2008-12-21; First posted 2008-12-23 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Osteochondritis of the Femoral Head
Keywords: Mesenchymal Stem Cells; Osteonecrosis of the Femoral Head
MeSH Terms: conditions — Legg-Calve-Perthes Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell (Experimental): mesenchymal stem cell infusion and bone marrow mononuclear cell infusion
  Interventions: Biological: mesenchymal stem cell infusion; Biological: bone marrow mononuclear cell infusion

INTERVENTIONS:
Biological: mesenchymal stem cell infusion
  Other Names: MSC infusion
Biological: bone marrow mononuclear cell infusion
  Other Names: BMMNC infusion

SUMMARY:
Mesenchymal Stem Cells (MSCs) have been shown to have immunosuppressive and repairing properties. Bone marrow mononuclear cells (BMMNCs) have revascularization properties and complimentary effects to MSCs. The investigators will infuse expanded autologous MSCs and BMMNCs into patients with osteonecrosis of the femoral head. The study purpose is to examine whether this treatment will result in improvement in osteonecrosis of the femoral head.

DETAILED DESCRIPTION:
Mesenchymal Stem Cells (MSCs) have been shown to have immunosuppressive and repairing properties. Bone marrow mononuclear cells (BMMNCs) have revascularization properties and complimentary effects to MSCs. Patients in this study will receive infusion of expanded autologous MSC and BMMNCs. The puncture of femoral artery will be conducted with digital subtraction angiography(DSA), and the tubes will be inserted into medial femoral circumflex artery,lateral femoral circumflex artery and obturatou artey. The study will evaluate the safety and effectiveness of MSC infusion in patients with osteonecrosis of the femoral head. This study will last for 5 years. Patients will undergo infusions at Day 0. Afterward, patients will be evaluated for response, and undergo X-ray examination, CT and MR scanning at a 6-month interval.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 12 to 60 years old.
* Association Research Circulation Osseous(ARCO) Classification criteria for osteonecrosis of the femoral head: ARCO phase I and phase II.
* Able to give informed consent.

Exclusion Criteria:

* Pregnant women.
* Previous history of malignancy
* Active infection including hepatitis B, hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB.
* Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in the past 6 months.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* Any illness that in the opinion of the investigator would jeopardize the ability of the Patient to tolerate this treatment.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The femoral head blood-supply artery angiographies and the areas of femoral head necrosis | 2

SECONDARY OUTCOMES:
Coxa joint paining | 2
Walking distance | 2
Joint functions | 2
Life | 2

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, professor, Principal Investigator — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China